CLINICAL TRIAL: NCT00376194
Title: An Investigation of the Efficacy of Mercury Chelation as a Treatment for Autism Spectrum Disorder
Brief Title: Mercury Chelation to Treat Autism
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 060238; 06-M-0238
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Autism; Asperger's Disorder; Child Development Disorders, Pervasive
Keywords: Pervasive Developmental Disorder; Alternative Therapy; Autism; Asperger's Disorder; Clinical Trial; Autism Spectrum Disorder; ASD; Asperger Disorder
MeSH Terms: conditions — Autistic Disorder; Asperger Syndrome; Child Development Disorders, Pervasive; Autism Spectrum Disorder | interventions — Succimer

INTERVENTIONS:
Drug: DMSA

SUMMARY:
This study will examine whether DMSA, an oral chelating agent that removes mercury and other metals from the body, is beneficial for children with autism. DMSA is commonly used to treat autism, although it has never been tested in a controlled study and there is no proof that it helps children with the disorder. Support for its use is based on single-case reports of benefits of chelation with DMSA. This study will help determine whether or not DMSA is useful for treating autism.

Children between 4 and 10 years of age with autism spectrum disorder who weigh at least 33 pounds, who have detectable, but not toxic, levels of mercury or lead in the blood, and who have not previously received chelation therapy may be eligible for this study.

Participants complete a medical history, behavioral and psychological assessment and physical examination. Blood, hair, urine and stool samples are collected for testing.

Because DMSA can remove minerals the body needs, such as zinc and iron, as well as the toxic lead and mercury, participants take a daily multivitamin supplement starting 1 month before beginning chelation therapy and continuing for the duration of treatment. After 1 month of the supplementation regimen, the children are assigned to receive DMSA or placebo for 12 weeks, divided into six 2-week cycles. They take the assigned drug 3 times a day on days 1, 2 and 3 of each cycle and continue the multivitamin every day.

The children are seen in the clinic immediately before and after the first, third and sixth cycles. At each checkup, the parent or guardian answers a set of questions about the child's autism symptoms, physical health and medication side effects. Blood, urine and stool samples are collected for laboratory testing.

...

DETAILED DESCRIPTION:
Chelation of metals is widely used in the community to treat individuals with Autism Spectrum Disorder (ASD), with some surveys estimating that 1 in 12 children with autism have undergone chelation. This widespread use reflects the hypothesis that many cases of ASD are caused by exposure to thimerosal, an ethylmercury-based compound used previously in the US as a vaccine preservative for routine childhood immunizations. The prevalent use of chelation therapy stands in stark contrast with the lack of scientific or clinical evidence of efficacy, and creates a public health imperative for empiric data. Thus we propose a controlled trial of the effects of chelation on the core behavioral symptoms and overall functioning of children with ASD. The present investigation is a double-blind, randomized placebo-controlled study of the oral chelating agent meso-2,3-dimercaptosuccinic acid (DMSA; succimer) among 120 children, ages four to ten years, who meet criteria for ASD. Pre- and post-treatment behavioral ratings will be used to evaluate the efficacy of chelation. In addition, children will undergo comprehensive medical history, physical examination and laboratory analyses.

Our objective is to quantify differences in behavioral functioning between the chelation treatment group and the placebo control group. Analysis of mercury levels before and during the course of treatment will be used to confirm the expected DMSA-induced excretion of mercury and to identify differences among children in the extent of excretion. Our primary hypothesis is that, on average and relative to the control group, children with ASD who undergo chelation with DMSA will show greater improvements in communication and social behavior.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects may be included in the study only if they meet all of the following criteria:

* Male or female subjects, four to ten years of age.
* Meets research criteria for ASD (specifically, autism, Asperger Disorder, or Pervasive Developmental Disorder - Not Otherwise Specified).
* Detectable (greater than 0.1 microgram per deciliter) levels of blood lead and/or blood mercury.
* Each legal guardian must have a level of understanding sufficient to agree to all required tests and examinations. Each legal guardian must understand the nature of the study and must provide written consent to study protocol.

EXCLUSION CRITERIA:

* History of allergic reaction to sulfur or thiol-containing substances
* History of previous chelation therapy for autism
* History of uncontrolled epilepsy
* Weight less than 15 kg at screening
* Presence of a chronic medical condition that might interfere with study participation in which study participation would be contraindicated or in which there may be clinically significant abnormal baseline laboratory results.
* Level of lead above 10 microgram per d, or level of mercury over 44 microgram per deciliter (toxic levels that require intervention with chelation and preclude placebo assignment) or other evidence of heavy metal toxicity.
* Recent (less than two months prior to study entry) initiation of behavior therapy

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2006-09; Study Completion 2007-03

PRIMARY OUTCOMES:
Improvement in social reciprocity.

SECONDARY OUTCOMES:
Improvement in language skills, decrease in blood mercury levels.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Aposhian HV, Aposhian MM. meso-2,3-Dimercaptosuccinic acid: chemical, pharmacological and toxicological properties of an orally effective metal chelating agent. Annu Rev Pharmacol Toxicol. 1990;30:279-306. doi: 10.1146/annurev.pa.30.040190.001431. PMID 2160791
- [Background] Bernard S, Enayati A, Redwood L, Roger H, Binstock T. Autism: a novel form of mercury poisoning. Med Hypotheses. 2001 Apr;56(4):462-71. doi: 10.1054/mehy.2000.1281. PMID 11339848
- [Background] Chisolm JJ Jr. Safety and efficacy of meso-2,3-dimercaptosuccinic acid (DMSA) in children with elevated blood lead concentrations. J Toxicol Clin Toxicol. 2000;38(4):365-75. doi: 10.1081/clt-100100945. PMID 10930052